CLINICAL TRIAL: NCT04765124
Title: A Multicenter Chart Review Study for Evaluating The Efficacy and Safety of Neoadjuvant Trastuzumab Plus Taxane With and Without Pertuzumab Therapy in Locally Advanced HER2 Positive Breast Cancer Patients
Brief Title: The Efficacy and Safety of Neoadjuvant Trastuzumab Plus Taxane With and Without Pertuzumab Therapy
Acronym: HER2PATH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahmet Bilici (Other)
Collaborators: Medipol University (Other); Bezmialem Vakif University (Other); Koç University (Other); Medical Park AG (Industry); Uludag University (Other); Akdeniz University (Other); Dicle University (Other); Trakya University (Other); Ankara City Hospital Bilkent (Other); Memorial Ankara Hospital (Other); Gulhane Training and Research Hospital (Other Government); Liv Hospital Ankara (Other); Ankara University (Other); Istanbul Medeniyet University (Other); Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other); Acıbadem Atunizade Hospital (Other); Inonu University (Other); Ege University (Other)
Responsible Party: Sponsor-Investigator, Ahmet Bilici, Prof., Medipol University
Organization: Medipol University (Other)
Other Study IDs: ML42876
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a Non-Interventional Study (NIS) with secondary data usage. It is designed as a multi-center retrospective cohort study in which the data of adult locally advanced HER2-positive breast cancer patients, who are treated with as neoadjuvant therapy, who underwent breast surgery in participating centers, were taken from hospital records.

The source population is academic or community oncology centers treating patients with breast cancer from Turkey.

The study population is planned to be the subgroup of breast cancer patients, who are treated with trastuzumab plus taxane with or without pertuzumab as neoadjuvant therapy, and underwent breast surgery at the participating centers.

The study is anticipated to include approximately 1500 patients from 20 sites.

DETAILED DESCRIPTION:
In 2013, the Food and Drug Agency (FDA) granted accelerated approval to pertuzumab for use in the neoadjuvant setting with trastuzumab and chemotherapy for HER2+ locally advanced breast cancer (either greater than 2 cm in diameter or node positive), based on improvement in pCR in the NeoSphere (Neoadjuvant Study of Pertuzumab and Herceptin in an Early Regimen Evaluation) and TRYPHAENA (Trastuzumab plus Pertuzumab in Neoadjuvant HER2- positive Breast Cancer) studies. Full approval of pertuzumab in the early stage for patients at high risk of recurrence was recently received based on results of the adjuvant APHINITY study. NeoSphere study demonstrated a higher breast pCR rate with THP 17 (docetaxel, trastuzumab, pertuzumab) as compared to TH (breast pCR 45.8 versus 29%), and TRYPHAENA study also demonstrated high total pCR rates with FEC (5- fluorouracil, epirubicin, and cyclophosphamide)-THP (pCR 54.7%) and TCHP (docetaxel, carboplatin, HP, pCR 63.6%).

Pertuzumab is a humanized monoclonal antibody and is the first of a novel class of HER2-targeted agents known as HER2 dimerization inhibitors. This agent bind to a distinct epitope on the extracellular domain of the HER2 receptor (the domain II dimerization arm), blocking the interaction between HER2 and other HER family receptors. Potent inhibition of HER-mediated intracellular signaling results in cancer cell growth inhibition and death.

In Turkey, Pertuzumab has been authorized as neoadjuvant therapy for breast cancer patients since March 2019. Before this date pertuzumab was also available after patient- based approvals. Due to lack of local data regarding outcomes of pertuzumab in neoadjuvant therapy for breast cancer patients, this study will be the first in this area, in terms of national real world data.

This study is a Non-Interventional Study (NIS) with secondary data usage. It is designed as a multi-center retrospective cohort study in which the data of adult breast cancer patients, who are treated with as neoadjuvant therapy and underwent breast surgery in participating centers, were taken from hospital records.

NIS secondary data use based on electronic health records and paper files. Required key, primary and secondary variables will be ready including pCR data at the hospital records. If not, at the time of surgery there will be biopsy / imaging and other laboratory results, so primary or sub-investigator could also assess response and note as a source document.

All patients' data planned to be collected in line with this study protocol after the ethics approval of the study.

This retrospective design and secondary data use will help to reach endpoints in a short time with a 1500 target patient number.

This study is planned to be performed on nation-wide across Turkey from 20 oncology clinics.

The data will be collected into the database via an electronic case report form (e-CRF). Principal investigators at each participating site will be in charge of transferring patient data into the e-CRF. Data from the initial diagnosis of each patient until the last requested and available data in the patient charts at each participating site will be collected.

The primary variables for this study are as follows:

Demographics Clinical Information Diagnosis date Clinical Stage Pathological stage(TNM stage) Receptor status Histologic subtype Imaging details Neoadjuvant therapy Start date Stop date Response at the time of surgery Imaging after neoadjuvant treatment if available Recurrence if available Breast surgery Surgery type Operation date Imaging after operation Adjuvant therapy Start date Stop date Response Patients status (Ex, alive, last follow-up date,lost to follow-up)

Secondary Variables

The secondary variables for this study are as follows:

Adverse Events Incidence Therapy relationship Grade according to CTCAE Start/End date Outcomes : Hospitalization, intervention, ex, etc Recurrence date, death date if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years old and over
* Patients diagnosed as histologically confirmed (IHC score of 3+ and/or positive by ISH) locally advanced HER2-positive breast cancer with breast surgery.
* Patients who received as neoadjuvant therapy.

Exclusion Criteria:

* Patients transferred from an other hospital should not be included, however, patients' data transferred to an other hospital will be collected till transfer time

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients diagnosed as breast cancer will be recruited
Study Population: The source population is academic or community oncology centers treating patients with breast cancer from Turkey.
  The study population is planned to be the subgroup of breast cancer patients, who are treated with trastuzumab plus taxane with or without pertuzumab as neoadjuvant therapy, and underwent breast surgery at the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate Pathologic Complete Response (pCR) rate | 8 months
  pCR is defined as the absence of residual invasive disease on H&E evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0 in the current American Joint Committee on Cancer (AJCC) staging system).

SECONDARY OUTCOMES:
To evaluate 2 year Event-Free Survival (EFS) | 24 months
  2 year EFS events are defined from trastuzumab initiation as the first occurrence of one of; progression of disease that precludes surgery, local or distant recurrence or death to any cause in two years.
To evaluate 2-year Invasive Disease-Free Survival (IDFS) | 24 months
  IDFS, defined from trastuzumab initiation as absence of all of the following in two years; Ipsilateral invasive breast cancer recurrence, regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer, or second non-breast invasive cancer (Note: In-situ events are not included)
To evaluate the safety of trastuzumab plus taxane with or without pertuzumab in terms of grade 3, 4 and 5 according to CTCAE v.5.0 | 8 months
  Adverse events only grade 3 (severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care),4 (life-threatening consequences; urgent intervention indicated) and 5 (death related to AE) according to CTCAE v.5.0 will be collected. Adverse events will be listed as percentage according to system organ class and term

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Bilici, Prof, Principal Investigator — Medipol University Hospital
Locations (1):
- Medipol University Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No